CLINICAL TRIAL: NCT03600597
Title: Construct Validity and Reliability of the Selective Control of the Upper Extremity Scale in Children With Cerebral Palsy
Brief Title: Construct Validity and Reliability SCUES
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Research assistant, Gazi University
Other Study IDs: 77082166-302.08.01-
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy; Upper Extremity Dysfunction
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to determine construct validity, discriminant validity and intra- and interrater reliability of the Selective Control of the Upper Extremity Scale (SCUES).

DETAILED DESCRIPTION:
This study included children diagnosed with unilateral cerebral palsy. Children's upper extremity-selective motor controls were evaluated by video recording. Manual Ability Classification System and Taylor Hand Function Test were used to determine upper extremity functions

ELIGIBILITY:
Inclusion Criteria:

* Ages between 3-18 years
* Diagnosed as Cerebral Palsy (Hemiplegia)

Exclusion Criteria:

* Participants with an unstable situation regarding their tonus-regulating medications
* Participants had a botulinum toxin injection within the last 6 months, or any surgical correction within the last year

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with Unilateral Cerebral Play
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Selective Control of the Extremity Scale | 10 minutes
  SCUES administration required patients to perform specific isolated movement patterns at the shoulder (abduction/adduction), elbow (flexion/extension), forearm (supination/pronation), wrist (flexion/extension), and fingers/ thumb (grasp/release). Presence of mirror movements, movement of additional joints and motion less than available ROM are graded for movement at each joint level. Motion at each of the five joint levels is graded on a four-point scale: no SMC, moderately diminished SMC, mildly diminished SMC, and normal SMC.

SECONDARY OUTCOMES:
Jebsen Taylor Hand Function Test | 20 minutes
  The JTT measures movement, speed and manual dexterity. The subtests to assess hand function included turning over cards, simulated feeding, picking up small common objects, stacking checkers, picking up large objects, and picking up large heavy objects. Each task completion time was limited to 2 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Study Chair — Study chair
Locations (1):
- Gazi University, Ankara, Yeni̇mahalle, Turkey (Türkiye)